CLINICAL TRIAL: NCT01505907
Title: Phase I, Randomized, Double-Blind, Placebo Controlled, Dose Escalation,Single Dose, Safety, Tolerance, and Pharmacokinetic Study of CXB909 in Healthy Male Volunteers
Brief Title: Pharmacokinetic Study of CXB909 in Healthy Male Subjects
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CeNeRx BioPharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple
Other Study IDs: CXB909-100
Record Dates: First submitted 2012-01-05; First posted 2012-01-09 (Estimated); Last update posted 2012-01-09 (Estimated); Status verified 2012-01

CONDITIONS: Healthy
Keywords: Pharmacokinetics; Safety; Healthy Males

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- CXB909 15mg (Experimental): CXB909 15mg
  Interventions: Drug: CXB909
- CXB909 30mg (Experimental)
  Interventions: Drug: CXB909
- CXB909 60mg (Experimental)
  Interventions: Drug: CXB909
- CXB909 120mg (Experimental): Dose
  Interventions: Drug: CXB909
- CXB909 250mg (Experimental)
  Interventions: Drug: CXB909

INTERVENTIONS:
Drug: CXB909 — CXB909

SUMMARY:
The primary objective of this dose escalation study is to examine the safety, tolerability, and pharmacokinetic properties of single-doses of CXB909, compared to placebo, in healthy male volunteers. This study may evaluate five (5) dose levels of CXB909; however, the number of dose levels, as well as the dosages, may be adjusted after evaluation of in-study analysis of the safety, tolerability, and pharmacokinetic data. This study will attempt to identify the maximum tolerated single dose of CXB909.

ELIGIBILITY:
Inclusion Criteria:

1. Male, 18 to 50 years of age.
2. Able to read, understand, and provide written/dated informed consent before screening in the study, and must be willing to comply with all study procedures.
3. In good general health as ascertained by thorough medical history, physical examination (PE)including measurement of supine and standing vital signs, clinical laboratory studies, and 12-lead electrocardiogram (EKG).
4. Body Mass Index (BMI) > 21 and < 30.
5. Willing and able to be confined to the clinical research unit as required by the protocol.

Exclusion Criteria:

1. Presence of a significant acute or chronic medical disorder that might complicate evaluation of the study drug such as:

   * Any cardiovascular or cardiac condition.
   * Supine SBP≥145 mmHg and/or DBP ≥90 mmHg at Screening.
   * Diabetes mellitus.
   * Malignancy and/or chemotherapy within two years of screening, other than basal cell carcinoma. Malignancies more than two years prior may not preclude participation; however, must be reviewed on a case-by-case basis by the CeNeRx BioPharma, Inc., medical monitor.
   * Known or suspected hypersensitivity to CXB909.
   * Any gastrointestinal disease or digestive disorder, neurological, pulmonary, hepatic, renal, hematologic, endocrine and/or metabolic disease or disorder.
2. Current or past psychiatric illness.
3. Use of any prescription medications within 14 days of study drug administration.
4. Use of any over-the-counter (OTC) medication within seven days of study drug administration (including herbal remedies).
5. History of substance abuse, including alcohol abuse as defined by DSM-IV criteria,within the past 12 months.
6. Current use of tobacco products or any nicotine-containing products (e.g., gum, patch)for the prior three months.
7. Consumption of alcohol or caffeine/xanthine-containing drinks or foods within 72 hours of dosing on Day 1 (including any type of wines, caffeinated or decaffeinated herbal tea, and grapefruit products (e.g., fresh, canned, or frozen), Seville oranges and pomelos).
8. Abnormal screening medical/physical examination, unless the abnormality is considered unlikely to be affected by study participation, or confound interpretation of safety data.
9. A clinically significant clinical laboratory or EKG abnormality at screening; includes any of the following: aspartate transaminase (AST), alanine transaminase (ALT), or alkaline phosphate (ALP) >2.0 x the upper limit of normal (ULN); total bilirubin >1.5 x the ULN;serum creatinine >1.5 x the ULN; blood urea nitrogen (BUN) >1.5 x the ULN; and thyroid stimulating hormone (TSH) and/or free thyroxine (T4) outside of the normal limits.
10. Test positive for: Urine cannabinoids, cocaine, amphetamines, barbiturates, opiates or benzodiazepines, serum alcohol, hepatitis B or C, or nicotine use.
11. HIV/AIDS.
12. Participation in a clinical investigation within the last 45 days of screening.
13. Any other condition which, in the investigator's opinion, may place the subject at greater than normal risk of developing complications.
14. Donation of any blood product (one pint or greater) within the previous eight weeks of screening.
15. Planning to donate any blood product within eight weeks of end of study.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic Parameters | 1 Week
  The PK parameters to be determined will include: Tmax, t1/2, Cmax, AUClast, AUCinf, Vd/F and CL/F.

SECONDARY OUTCOMES:
Safety | 1 Week
  Descriptive statistics will be reported for adverse events; systolic and diastolic blood pressures; pulse; the respiration rate; QTC, PR, and QRS intervals; and the laboratory parameters. QTC will be calculated using both the Bazett and Fridericia corrections.